CLINICAL TRIAL: NCT03401827
Title: The Effect of Gemcitabine Plus Nab-paclitaxel as Secondary Chemotherapy in Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1710-067-894
Record Dates: First submitted 2017-12-30; First posted 2018-01-17 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Adenocarcinoma; Chemotherapy Effect
Keywords: pancreatic cancer; second line chemotherapy; nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine + nab-paclitaxel (Experimental): Case with chemotherapy (Gemcitabine + nab-paclitaxel)
  Interventions: Drug: Chemotherapy (Gemcitabine + nab-paclitaxel)

INTERVENTIONS:
Drug: Chemotherapy (Gemcitabine + nab-paclitaxel) — Nanoparticle albumin-bound paclitaxel (125 mg/m2) miv over 30 min, Day 1,8,15
  Gemcitabine (1,000mg/m2) and N/S 150mL miv over 30 min, Day 1,8,15
  Other Names: GnP

SUMMARY:
Pancreatic cancer is a very poor prognosis and has a high mortality rate. The clinical results have improved somewhat with the combination therapy of chemotherapy as the first-line treatment. However, effective secondary chemotherapy after these first-line treatment failures is limited. Recently, FOLFIRINOX has been used in patients with locally advanced or metastatic pancreatic cancer who have good performance in Korea. Gemcitabine + nab-paclitaxel (GnP) as a second-line treatment after FOLFIRINOX may be expected to be considerable. The aim of this study was to evaluate the efficacy of GnP as a second-line treatment after failed FOLFIRINOX treatment for locally advanced or metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic cancer is a very poor prognosis and has a high mortality rate. It is not clear that the improvement of clinical outcome due to anticancer drugs is not clear compared to other carcinomas. In particular, the 5-year survival rate of metastatic pancreatic cancer is still only about 2%, and the clinical results have improved somewhat with the combination therapy of chemotherapy as the first-line treatment. However, effective secondary chemotherapy after these first-line treatment failures is limited. Meta-analysis has reported that life expectancy is significantly increased in patients receiving second-line chemotherapy after failure of primary chemotherapy. However, it is not yet clear which cancer treatment is most effective. In the NCCN guideline (ver. 2017.2), the second trial of chemotherapy for locally advanced or metastatic pancreatic cancer is the most recommended clinical trial.Recently, FOLFIRINOX has been used in patients with locally advanced or metastatic pancreatic cancer who have good performance in Korea. The response rate of the treatment is 30%, and many patients require secondary chemotherapy. In a practice guideline published by the American Society of Clinical Oncology, Gemcitabine + nab-paclitaxel(GnP) is the only recommended combination for patients failing primary treatment with FOLFIRINOX. In light of the results of previous reports, the efficacy of GnP as a second-line treatment after FOLFIRINOX may be expected to be considerable, but there is a lack of studies reporting GnP therapy on the second line after FOLFIRINOX failure as a first-line treatment. The aim of this study was to evaluate the efficacy of GnP as a second-line treatment after failed FOLFIRINOX treatment for locally advanced or metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
1. Inclusion criteria

   1. Patient whose age is 20 years or older
   2. ECOG Performance Status 0-2
   3. Pathologically confirmed pancreatic adenocarcinoma
   4. Patients with locally advanced or distant metastasis status
   5. Patients who had undergone primary chemotherapy with previous FOLFIRINOX and whose disease progress was confirmed
   6. Patients whose consent was obtained (non-insurance agreement)
2. Exclusion Criteria

   1. Those who can not obtain consent
   2. Those who refuse chemotherapy
   3. ECOG Performance Status 3 or higher
   4. Multiple organ failure is accompanied
   5. Severe comorbidities other than cancer that do not expect a sufficient survival period over 1 month
   6. Allergy to the test drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
survival rate | 6 months
  survival rate at 6 months after 2nd line chemotherapy

SECONDARY OUTCOMES:
overall survival | till death or follow-up loss or end of study up to 2 years
  overall survival after 2nd line chemotherapy
Progression free survival | till death or follow-up loss or end of study up to 2 years
  duration till progression after 2nd line chemotherapy
Disease control rate | 6 months
  SD (stable disease) + PR (partial response) + CR (complete response) after 2nd line chemotherapy
adverse event | till death or follow-up loss or end of study up to 2 years
  all reported adverse events after 2nd line chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, MD, Ph.D, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Huh G, Lee HS, Choi JH, Lee SH, Paik WH, Ryu JK, Kim YT, Bang S, Lee ES. Gemcitabine plus Nab-paclitaxel as a second-line treatment following FOLFIRINOX failure in advanced pancreatic cancer: a multicenter, single-arm, open-label, phase 2 trial. Ther Adv Med Oncol. 2021 Nov 10;13:17588359211056179. doi: 10.1177/17588359211056179. eCollection 2021. PMID 34790261